CLINICAL TRIAL: NCT02352831
Title: Phase I/II Study Combining Tosedostat With Capecitabine in Patients With Metastatic Pancreatic Adenocarcinoma
Brief Title: Tosedostat With Capecitabine in Patients With Metastatic Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient funding and drug supply from manufacturer
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201503074
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Pancreatic Cancer; Cancer of Pancreas; Cancer of the Pancreas; Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — tosedostat; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I (tosedostat + capecitabine) (Experimental): * The phase I study will be conducted in the standard 6-patient-per-cohort dose de-escalation fashion.
  * Tosedostat by mouth daily Days 1-21 of each 21-day cycle. Dose Level 0 (starting dose) = 120 mg PO daily and Dose Level -1 = 60 mg PO daily. All 6 patients in the Phase 1 received 120 mg starting dose of tosedostat.
  * Capecitabine 1000 mg/m^2 by mouth BID Days 1-14 of each 21-day cycle
  * Fresh tissue biopsy: Patients who have a partial response at the end of cycle 2 will be required to undergo biopsy if deemed safe for the patient and tissue is feasible to obtain.
  Interventions: Drug: Tosedostat; Drug: Capecitabine; Procedure: Fresh tissue biopsy
- Phase II (tosedostat + capecitabine) (Experimental): * Tosedostat (dose determined by Phase I portion of study) by mouth daily Days 1-21 of each 21-day cycle
  * Capecitabine by mouth BID Days 1-14 of each 21-day cycle
  Interventions: Drug: Tosedostat; Drug: Capecitabine; Procedure: Fresh tissue biopsy

INTERVENTIONS:
Drug: Tosedostat
Drug: Capecitabine
  Other Names: Xeloda
Procedure: Fresh tissue biopsy — Patients who have a partial response at the end of cycle 2 will be required to undergo biopsy if deemed safe for the patient and tissue is feasible to obtain.

SUMMARY:
There are two parts to this study: the goal of the first part of the study is to find the best dose of tosedostat when given in combination with capecitabine. The goal of the second part of the study is to look at how participants respond to treatment with tosedostat and capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven metastatic or inoperable pancreatic adenocarcinoma.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm with CT scan or MRI, as >20 mm by chest x-ray, or >10 mm with calipers by clinical exam.
* Must have progressed on, been intolerant to, or refused gemcitabine-based therapy.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,000/mcl
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ 2.0 mg/dL
  * Creatinine ≤ 2.0 mg/dL
  * AST or ALT ≤2.5 IULN (≤5X IULN if liver metastases are present)
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Chemotherapy < 2 weeks prior to the first planned dose of study treatment.
* Radiotherapy < 3 weeks prior to the first planned dose of study treatment.
* A history of other malignancy ≤ 2 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Currently receiving any other investigational agents.
* Known brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to tosedostat or capecitabine or other agents used in the study.
* Previous treatment with any aminopeptidase inhibitor.
* Previous exposure to either 5-FU or capecitabine at a systemic dose except for use in concurrent chemoradiation.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency or severe renal impairment (creatinine clearance < 30 mL/min by Cockcroft-Gault formula), as this would preclude use of capecitabine.
* Significant cardiovascular disease defined as:

  * Myocardial infarction within 6 months of screening.
  * Unstable angina pectoris
  * Uncontrolled or clinically significant arrhythmia Grade ≥ 2
  * LVEF ≤ below institutional limits at screening
  * Congestive heart failure NYHA class III or IV
  * Presence of clinically significant valvular heart disease
  * Baseline troponin I or T > IULN and b-type natriuretic peptide > IULN.
* Prior exposure to cardiotoxic agent, such as anthracyclines, within 3 months of enrollment.
* Patient must have a QTc interval on ECG ≤ 0.48 seconds by Bazett's calculation at screening.
* Patient may not be taking any drugs that prolong the QT/QTc interval. If patient is on any of these drugs, patient may enroll in the study if the drugs can be discontinued for at least 5 half-lives prior to the first dose of tosedostat and capecitabine.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Patients that are of childbearing age must have a negative pregnancy test at screening and agree on using contraception during the duration of the study.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with tosedostat or capecitabine. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2018-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Wang-Gillam, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 08/31/2015 and closed to participant enrollment on 12/22/2017.
Groups:
- Phase II (Tosedostat + Capecitabine): * Tosedostat (dose determined by Phase I portion of study) by mouth daily Days 1-21 of each 21-day cycle
  * Capecitabine by mouth BID Days 1-14 of each 21-day cycle
  * Fresh tissue biopsy: Patients who have a partial response at the end of cycle 2 will be required to undergo biopsy if deemed safe for the patient and tissue is feasible to obtain.
Period: Overall Study
Arm/Group | Phase I (Tosedostat + Capecitabine) | Phase II (Tosedostat + Capecitabine)
Started | 6 | 10
Completed | 6 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I (Tosedostat + Capecitabine) | Phase II (Tosedostat + Capecitabine) | Total
Number analyzed (Participants) | 6 | 10 | 16
Age, Continuous [Median (Full Range); unit: years] | 60.5 [42 to 73] | 69.5 [51 to 76] | 66 [42 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 10 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 9 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 10 | 16
Baseline CA19-9 [Mean (Full Range); unit: U/mL] | 331.22 [1.00 to 1697.90] | 2061.73 [19.70 to 8803.00] | 1255 [1.00 to 8803.00]

OUTCOME MEASURES:

1. Primary Outcome: Phase I Only: Recommended Phase II Dose of Tosedostat
Description: The recommended phase 2 dose (RP2D) is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle. If 0 or 1 of 6 patients in Dose Level 1 experience DLT during the first cycle, Dose Level 1 will be presumed to be the RP2D.
  DLTs are followed through completion of the first cycle.
Time Frame: Completion of cycle 1 of all participants in Phase I portion of study (approximately 14 months)
Population: This outcome measure is for Phase I participants only.
Measure: Number; unit: mg daily
Arm/Group | Phase I (Tosedostat + Capecitabine) | Phase II (Tosedostat + Capecitabine)
Number analyzed (Participants) | 6 | 0
mg daily | 120 |

2. Primary Outcome: Phase I Only: Number of Participants Who Experience Dose-limiting Toxicities (DLTs)
Description: * Possibly/probably/definitely related to study treatment in 1st cycle (cyc)
    *Grade (Gr) 4 neutropenia >7 day, Febrile neutropenia of any duration with temperature ≥ 38.5 °C, Gr 4 anemia requires transfusion therapy on more than 2 occasions in 7 days, Gr 4 thrombocytopenia
  * Possibly/probably/definitely related gr. 3/4 non-hematologic toxicity that occurs 1st cyc with the following EXCEPTIONS:
    * Gr 3 nausea/vomiting/diarrhea/anorexia <72 hours that returns to Gr 1 prior to the start of cyc 2, Gr 3 hand-foot syndrome will only be considered a DLT for patients who have received 1 week of supportive care treatment with no improvement, Gr 3 fatigue that returns to Gr 1 prior to the start of cyc 2, Gr 3 flu-like symptoms <72 hours that returns to Gr 1 prior to start of cyc 2, Gr 3 arthralgia or myalgias <72 hours that return to Gr 1 prior to the start of cyc 2, Gr 3 potassium/phosphorus/magnesium that is asymptomatic or of non-clinical significance <72 hours, Gr 3 hypoalbuminemia
Time Frame: Completion of cycle 1 of all participants in Phase I portion of study (approximately 14 months)
Population: This outcome measure is for Phase I participants only.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (Tosedostat + Capecitabine) | Phase II (Tosedostat + Capecitabine)
Number analyzed (Participants) | 6 | 0
Participants | 1 |

3. Primary Outcome: Progression-free Survival (PFS) Rate
Description: * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive disease (PD)
    * Target lesions: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
    * Non target lesions: Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Phase I and Phase II Combined: * Tosedostat by mouth daily Days 1-21 of each 21-day cycle
  * Capecitabine by mouth BID Days 1-14 of each 21-day cycle
  * Fresh tissue biopsy: Patients who have a partial response at the end of cycle 2 will be required to undergo biopsy if deemed safe for the patient and tissue is feasible to obtain.
Arm/Group | Phase I (Tosedostat + Capecitabine) | Phase II (Tosedostat + Capecitabine) | Phase I and Phase II Combined
Number analyzed (Participants) | 6 | 10 | 16
Participants | 3 | 8 | 11

4. Secondary Outcome: Overall Response Rate (ORR)
Description: * ORR = Complete response + partial response
  * Target lesions
    * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
    * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Non target lesions *Complete Response (CR): Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (Tosedostat + Capecitabine) | Phase II (Tosedostat + Capecitabine)
Number analyzed (Participants) | 6 | 10
Participants | 0 | 0

5. Secondary Outcome: Time-to-progression (TTP)
Description: -Progressive disease (PD)
  * Target lesions: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
  * Non target lesions: Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase
Time Frame: Up to 24 months
Measure: Median (Full Range); unit: days
Arm/Group | Phase I (Tosedostat + Capecitabine) | Phase II (Tosedostat + Capecitabine)
Number analyzed (Participants) | 6 | 10
days | 210.50 [44.00 to 681.00] | 94.50 [42.00 to 250.00]

6. Secondary Outcome: Overall Survival Rate (OS)
Time Frame: Up to 1 year from completion of treatment (median treatment length 81.50 days (28.00-346.00)
Measure: Count of Participants; unit: Participants
Groups:
- Phase I and Phase II (Tosedostat + Capecitabine): * Tosedostat by mouth daily Days 1-21 of each 21-day cycle
  * Capecitabine by mouth BID Days 1-14 of each 21-day cycle
Arm/Group | Phase I (Tosedostat + Capecitabine) | Phase II (Tosedostat + Capecitabine) | Phase I and Phase II (Tosedostat + Capecitabine)
Number analyzed (Participants) | 6 | 10 | 16
Participants | 3 | 2 | 5

7. Secondary Outcome: Number of Participants With a CA19-9 Response
Description: * CA19-9 is a tumor marker that is used in the management of pancreatic cancer. Rising CA19-9 levels may mean the tumor is growing and decreasing CA19-9 levels may mean the tumor is shrinking or the amount of cancer in the body is decreasing
  * A CA19-9 response means that the tumor marker has decreased over baseline (before treatment started) levels
Time Frame: Completion of treatment (median treatment length 81.50 days (28.00-346.00)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (Tosedostat + Capecitabine) | Phase II (Tosedostat + Capecitabine)
Number analyzed (Participants) | 6 | 10
Participants | 6 | 10

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality were collected from baseline through 30 days after treatment ended.
Arm/Group | Phase I (Tosedostat + Capecitabine) | Phase II (Tosedostat + Capecitabine)
All-Cause Mortality (participants affected / at risk) | 1/6 | 1/10
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/10
Other Adverse Events (participants affected / at risk) | 6/6 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I (Tosedostat + Capecitabine) (N=6) | Phase II (Tosedostat + Capecitabine) (N=10)
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Colon obstruction (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Superficial thrombephemelebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I (Tosedostat + Capecitabine) (N=6) | Phase II (Tosedostat + Capecitabine) (N=10)
Anemia (Blood and lymphatic system disorders) | 1 | 2
Blurred vision (Eye disorders) | 0 | 2
Dry eye (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Mucositis-oral (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Edema limbs (General disorders) | 2 | 3
Fatigue (General disorders) | 3 | 1
Fever (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Sensation to cold (General disorders) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Toe infection (Infections and infestations) | 1 | 0
Alkaline phosphatase (Investigations) | 0 | 4
Blood bilirubin increased (Investigations) | 0 | 1
Creatinine increase (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 4
Hemoglobin decrease (Investigations) | 6 | 6
Hypocalcemia (Investigations) | 0 | 2
Increased amylase (Investigations) | 0 | 1
Increased lipase (Investigations) | 0 | 1
Lymphocytes decrease (Investigations) | 2 | 4
Neutrophil count decrease (Investigations) | 1 | 0
Platelet count decrease (Investigations) | 6 | 5
White blood cells decrease (Investigations) | 2 | 3
aPTT increase (Investigations) | 0 | 1
ALT increase (Metabolism and nutrition disorders) | 3 | 3
AST increase (Metabolism and nutrition disorders) | 3 | 3
Anorexia (Metabolism and nutrition disorders) | 3 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Tingling of lips (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT02352831/Prot_SAP_000.pdf